CLINICAL TRIAL: NCT06698575
Title: A Phase 1a/1b, Blinded, Placebo-Controlled Study of the Safety, Tolerability and Pharmacokinetics of Single- and Multiple Ascending Doses of ABI-1179 in Healthy Subjects and in Subjects Who Are Seropositive for Herpes Simplex Virus Type 2 With Recurrent Genital Herpes
Brief Title: A Study to Assess the Safety, Pharmacokinetics, and Tolerability of ABI-1179 in Healthy Subjects and in Subjects Seropositive for HSV-2 With Recurrent Genital Herpes
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABI-1179-101
Record Dates: First submitted 2024-11-08; First posted 2024-11-21 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Genital Herpes Simplex Type 2
Keywords: ABI-1179, PK, Healthy Participants, HSV-2, Recurrent Genital Herpes
MeSH Terms: conditions — Herpes Genitalis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: SAD Cohorts 1-5, ABI-1179 (Experimental): Single dose of ABI-1179 (tablet) in Part A for cohorts 1-5
  Interventions: Drug: ABI-1179; Drug: ABI-1179 Placebo
- Part A:SAD Cohorts 1-5, Placebo (Placebo Comparator): Single dose of matching placebo (tablet) in Part A for Cohorts 1-5
  Interventions: Drug: ABI-1179; Drug: ABI-1179 Placebo
- Part A: (SAD) Fed Cohort 6 or 7, ABI-1179 (Experimental): Single dose of ABI-1179 (tablet) in Part A for Cohort 6 or 7, food effect
  Interventions: Drug: ABI-1179; Drug: ABI-1179 Placebo
- Part B: MAD Cohorts 1-4, ABI-1179 (Experimental): Weekly dose ofABI-1179 (tablet) in Part B for Cohorts 1-4. May have loading dose.
  Interventions: Drug: ABI-1179; Drug: ABI-1179 Placebo
- Part B: MAD Cohorts 1-4 Placebo (Placebo Comparator): Weekly dose of matching placebo (tablet) in Part B for Cohorts 1-4.
  Interventions: Drug: ABI-1179; Drug: ABI-1179 Placebo

INTERVENTIONS:
Drug: ABI-1179 — Once daily tablet dosing (SAD), or weekly tablet dosing over 29 days (MAD)
Drug: ABI-1179 Placebo — Once daily tablet dosing (SAD), or weekly tablet dosing over 29 days (MAD)

SUMMARY:
This study is designed to assess safety, tolerability, and pharmacokinetics (PK) of single ascending dose (SAD) of ABI-1179 in Part A in healthy participants and multiple-ascending doses (MAD) of ABI-1179 in Part B in participants seropositive for Herpes Simplex Virus Type 2 (HSV-2) with recurrent genital herpes. Effect of food will also be evaluated in Part A.

ELIGIBILITY:
Part A: Inclusion Criteria:

* Subject has a body mass index (BMI) between ≥18.0 and <32.0 kg/m2
* In good health (as determined by the Investigator) based on medical history, physical examination, ECG, and clinical laboratory results.
* Female subjects must be non-pregnant and have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Day-1 or Day 1 (predose).
* Agreement to comply with protocol-specified contraceptive requirements.

Part B: Inclusion Criteria:

* Subject has a body mass index (BMI) between ≥18.0 and <32.0 kg/m2
* Other than HSV infection, is in good health (as determined by the investigator) based on medical history, physical examination, ECG, and clinical laboratory results.
* Female subjects must be non-pregnant and have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Day 1 (predose).
* Agreement to comply with protocol-specified contraceptive requirements

Part A and B: Exclusion Criteria:

* Current infection of human immunodeficiency virus (HIV), hepatitis B virus, (HBV), hepatitis C virus (HCV), acute hepatitis A virus (HAV), or acute hepatitis E virus (HEV).
* History of any illness that, in the opinion of the Investigator, might confound the results of the study, pose an additional risk in administering study drug to the subject, or condition known to interfere with the absorption /distribution/ elimination of drugs.
* History of any significant drug-related allergic reactions such as anaphylaxis, Stevens-Johnson Syndrome, urticaria, or multiple drug allergies.
* History of persistent alcohol abuse or illicit drug abuse within 3 years prior to screening.
* Has participated in a clinical study involving administration of either an investigational or a marketed drug within 30 days or 5 half-lives before screening, whatever is longer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2024-12-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Time Curve, (AUC) of ABI-1179 | SAD Cohorts: before and at pre-specified timepoints up to 144 hours after dosing. MAD Cohorts: before and at pre-specified time points up to 8 hours after dosing.
Maximum Observed Plasma Concentration (Cmax) of ABI-1179 | SAD Cohorts: before and at pre-specified timepoints up to 144 hours after dosing. MAD Cohorts: before and at pre-specified time points up to 8 hours after dosing.
Time to Cmax (Tmax) of ABI-1179 | SAD Cohorts: before and at pre-specified timepoints up to 144 hours after dosing. MAD Cohorts: before and at pre-specified time points up to 8 hours after dosing.
Apparent Terminal Elimination Half Life ( t 1/2) ABI-1179 | SAD Cohorts: before and at pre-specified timepoints up to 144 hours after dosing. MAD Cohorts: before and at pre-specified time points up to 8 hours after dosing.
Apparent Systemic Clearance (CL/F) of ABI-1179 | SAD Cohorts: before and at pre-specified timepoints up to 144 hours after dosing. MAD Cohorts: before and at pre-specified time points up to 8 hours after dosing.
Apparent Volume of Distribution (Vz/F) of ABI-1179 | SAD Cohorts: before and at pre-specified timepoints up to 144 hours after dosing. MAD Cohorts: before and at pre-specified time points up to 8 hours after dosing.
Dose normalized AUCs and Cmax of ABI-1179 | SAD Cohorts: before and at pre-specified timepoints up to 144 hours after dosing. MAD Cohorts: before and at pre-specified time points up to 8 hours after dosing.
Proportion of subjects with adverse events (AEs), premature treatment discontinuation due to AE's and abnormal laboratory results. | Up to 56 days after last dose.

SECONDARY OUTCOMES:
SAD Cohorts: Comparison of Plasma AUC between fasted and fed treatments | MAD Cohorts: At pre-specified time points from Days 8 to 36.
SAD Cohorts: Comparison of plasma Cmax between fasted and fed treatments | SAD Cohorts: before and at pre-specified timepoints up to 144 hours after dosing.
MAD Cohort: If applicable comparison of plasma AUC and Cmax with and without loading doses | MAD Cohorts At pre-specified timepoints from Days 8 to 36
MAD Cohorts: Difference in viral shedding rate (number of anogenital swabs positive for HSV-2 DNA/total number of swabs) across treatments. | MAD Cohorts: At pre-specified time points from Days 8 to 36.
MAD Cohorts: in mean and median HSV-2 DNA copies/ml for swab samples positive for HSV-2 DNA across treatments | MAD Cohorts: At pre-specified time points from Days 8 to 36.
MAD Cohorts: Difference in the proportion of swab samples with HSV-2 DNA>4log10 copies/mL across treatments (number of swabbing samples with HSV-2 DNA >4 log10 copies/mL / total number of swabs obtained). | MAD Cohorts: At pre-specified time points from Days 8 to 36.
MAD Cohorts: Difference in number of shedding episodes during the swabbing period across treatments. | MAD Cohorts: At pre-specified time points from Days 8 to 36.
MAD Cohorts: Difference in duration of shedding episodes during the swabbing period across treatments. | MAD Cohorts: At pre-specified time points from Days 8 to 36.
MAD Cohorts: Difference in the subclinical shedding rate (number of swabs positive for HSV-2 DNA in the absence of lesions/total number of swabs in the absence of lesions) across treatments. | MAD Cohorts: At pre-specified time points from Days 8 to 36.
MAD Cohorts: Difference in the lesion rate during the swabbing period across treatments. | MAD Cohorts: At pre-specified time points from Days 8 to 36.
MAD Cohorts: Difference in lesion duration during the swabbing period across treatments | MAD Cohorts: At pre-specified time points from Days 8 to 36.
MAD Cohorts: Difference in the recurrence rate (number of reappearances of lesions during the swabbing period/total days assessed) across treatments. | MAD Cohorts: At pre-specified time points from Days 8 to 36.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (4):
  - Alliance for Multispecialty Research, Kansas City, Missouri
  - Rochester Clinical Research, Rochester, New York
  - Seattle Clinical Research Center, Seattle, Washington
  - University of Washington Virology Research Clinic, Seattle, Washington
- Australia (6):
  - East Sydney Doctors, Darlinghurst, Australia
  - Royal Melbourne Hospital, Parkville, Australia
  - Taylor Square Private Clinic, Surry Hills, Australia
  - Momentum Clinical Research, Sydney, Australia
  - Canopy Clinical Wollongong, Wollongong, Australia
  - Momentum Sunshine, Melbourne, Au
- New Zealand (8):
  - New Zealand Clinical Research, Auckland, New Zealand
  - New Zealand Clinical Research, Christchurch, New Zealand
  - Pacific Clinical Research Network, Nelson, New Zealand
  - Momentum Palmerston North, Palmerston North, New Zealand
  - Pacific Clinical Research Network, Rotorua, New Zealand
  - Pacific Clinical Research Network, Upper Hutt, New Zealand
  - Momentum Kapiti, Waikanae, New Zealand
  - Pacific Clinical Research Network, Hamilton, New